CLINICAL TRIAL: NCT03221777
Title: Atrial Fibrillation Occurring Transiently With Stress (AFOTS): Understanding the Risks of Recurrent AF. Study in Non-cardiac Surgery and in Medical Illness Patients.
Brief Title: Atrial Fibrillation Occurring Transiently With Stress (AFOTS)
Acronym: AFOTS
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Cardiovascular Society (Other); Canadian Stroke Prevention Intervention Network (Other)
Responsible Party: Principal Investigator, William McIntyre, Research Fellow, Population Health Research Institute
Other Study IDs: AFOTS
Record Dates: First submitted 2017-06-30; First posted 2017-07-19 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation New Onset

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- AFOTS - Medical Illness Cases: Patients who have AF detected for the first time in the setting of an acute non-cardiovascular medical (i.e. non-surgical ).
  14 day patch ECG monitor at 1 month and 6 months after hospital discharge
  Interventions: Diagnostic Test: 14 Day ECG Patch (Zio XT Patch, iRhythm Technologies)
- Medical Illness Controls: Patients without a history of AF who are hospitalized for an acute non-cardiovascular medical (i.e. non-surgical) and do not have AF detected.
  14 day patch ECG monitor at 1 month and 6 months after hospital discharge
  Interventions: Diagnostic Test: 14 Day ECG Patch (Zio XT Patch, iRhythm Technologies)
- AFOTS - Non-cardiac surgery Cases: Patients who have AF detected for the first time following non-cardiac surgery.
  14 day patch ECG monitor at 1 month and 6 months after hospital discharge
  Interventions: Diagnostic Test: 14 Day ECG Patch (Zio XT Patch, iRhythm Technologies)
- Non-cardiac Surgery Controls: Patients without a history of AF who are hospitalized after non-cardiac surgery and do not have AF detected.
  14 day patch ECG monitor at 1 month and 6 months after hospital discharge
  Interventions: Diagnostic Test: 14 Day ECG Patch (Zio XT Patch, iRhythm Technologies)

INTERVENTIONS:
Diagnostic Test: 14 Day ECG Patch (Zio XT Patch, iRhythm Technologies) — The ZIO XT Patch (http://www.irhythmtech.com/zio-solution/zio-patch/) is an ultra-portable wearable adhesive patch monitor that provides continuous single-lead ECG recording for up to 14 days. It has been cleared by the FDA for arrhythmia detection and is in current clinical use in the U.S.[87]. It will be used in this study under an investigational testing authorization by Health Canada. The ZIO XT Patch is a single-use device worn over the left pectoral region with a skin adhesive (Figure 4). Its small, lightweight, water-resistant, patch-based design has advantages for patients compared with traditional ECG screening methods (e.g. Holter, event loop recorders, mobile outpatient telemetry systems), which are all more cumbersome and require detachable wired leads, two or more removable skin contact electrodes, plus separate recording units (+/- smartphone attachment).

SUMMARY:
Rationale Atrial fibrillation (AF) often occurs transiently in the setting of an acute stressor (e.g.

medical illness or surgery). Uncertainty exists as to whether AF Occurring Transiently with Stress (AFOTS) is secondary to a reversible precipitant and is benign, or is a first presentation of paroxysmal AF and associated with a risk of stroke. AFOTS is a common occurrence (>40% in some intensive care settings), but there is a lack of evidence to guide its management and guidelines have called for further research in this area. Retrospective data suggest that many patients with AFOTS (>50%) will experience recurrent AF. These estimates were obtained without using sensitive methods for AF detection, which raises the possibility that the true rate of recurrent AF is much higher. As the rate of recurrent AF increases, it becomes increasingly likely that AFOTS is just the first detection of typical "clinical" AF.

Objective To use a sensitive strategy to determine the rate of recurrent AF among patients who experienced AFOTS following i) non-cardiac surgery OR ii) medical illness, compared to matched controls.

Methods Two multi-centre, 138-patient, observational cohorts. AFOTS patients will have new AF, documented by 12-Lead ECG or surface monitoring, during hospitalization for non- cardiac surgery (Cohort 1) or medical illness (Cohort 2).

Controls will be patients without a history of AF who are matched for age (within 5 years), sex and exposure to stressor. Participants will wear a 14-day ECG monitor at 1 and 6 months after discharge. The endpoint is detection of AF.

Impact

If the incidence of AF after AFOTS is >80%, clinicians could be advised to treat AFOTS like "clinical" AF and initiate anticoagulation according to guidelines. Otherwise, a strategy of surveillance for AF would be advised.

Hypothesis

1. Patients who experience AFOTS will have a higher future incidence of AF and of stroke compared to patients exposed to a similar stressor but who did not develop AF.
2. The risk of recurrent AF after AFOTS will be sufficiently high (> 80%) to warrant routine initiation of long-term OAC in all cases.

ELIGIBILITY:
Inclusion Criteria:

Cases will be patients without a history of AF who experience new AFOTS during hospital admission for non-cardiac surgery (non-cardiac surgery study) OR medical illness (medical illness study) Controls will be patients who were exposed to a similar stressor but did not develop AF (matched for age within 5 years, sex and stressor).

All participants will have a CHA2DS2-VaSc score >1 for men, >2 for women.

Exclusion Criteria:

1. Documented prior history of AF.
2. Patients whose rhythm is AF at the time of discharge from hospital
3. Patients unsuitable for study follow-up because the patient:

   1. is unreliable concerning the follow-up schedule
   2. cannot be contacted by telephone
   3. has a life expectancy less than one year
4. Unwilling or unable to participate in the study
5. Presence of an implanted pacemaker or defibrillator.
6. Documented significant allergy to ECG electrode adhesive.
7. Residence in a chronic care facility
8. Diagnosed with Ischemic Stroke or Systemic embolism on admission
9. Primary cardiac admitting diagnosis (i.e. myocardial infarction, heart failure, pericarditis, arrhythmia)
10. Patients with Stage V Chronic Kidney Disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted for non-cardiac surgery OR medical Illness, who develop new Atrial Fibrillation Occurring Transiently With Stress (AFOTS) during hospital admission (case group), OR who are exposed to the same stressor, but did not develop AF (control group).
  All patients will be candidates for OAC therapy as per the Canadian Cardiovascular Society (CCS) AF algorithm [12]. Patients with a history of AF will be excluded from the study.
Sampling Method: Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation >/=30 s | 1 year

SECONDARY OUTCOMES:
Time to Atrial Fibrillation | 1 year
  Among AFOTS patients with the primary endpoint detected by the ECG patch monitor: time to first detection of AF >30 s.
Daily and total AF burden | 1 year
  Among AFOTS patients with the primary endpoint detected by the ECG patch monitor: daily and total AF burden.
Average duration per AF episode | 1 year
  Among AFOTS patients with the primary endpoint detected by the ECG patch monitor: average duration per AF episode
Other durations of Atrial Fibrillation | 1 year
  Among AFOTS patients, occurence of any AF episode lasting ≥30 seconds, ≥30 seconds to 5 minutes, >5 hours, and >24 hours (to facilitate comparison with other studies in the literature).( within 12 months post-enrolment)
Atrial Fibrillation at 1 and 6 months | 1 and 6 months
  Detection of the primary outcome at 1 and 6 months post enrolment.
Other clinical outcomes | 1 year
  Incidence of Clinical outcome events within 12 months post-enrolment (death, stroke, bleeding, embolism and hospitalization for heart failure or myocardial infarction), physician visits, hospitalizations and medication prescriptions.
OAC Use | 1 year
  Oral anticoagulant therapy use
Cost-effectiveness | 1 year
  Cost-effectiveness (cost per life year saved)
Cost-utility | 1 year
  cost-utility (cost per quality adjusted life year (QALY) gained) of AF screening
Patient adherence | 1 year
  Patient adherence with the monitoring devices (defined as the average number of monitoring days completed and reasons for non-adherence)
Patient satisfaction | 1 year
  patient satisfaction with the monitoring devices (as measured by user satisfaction surveys),
Sensitivity and Specificity | 1 year
  Estimated sensitivity, specificity of non-patch ECG monitoring(i.e. monitoring done outside of the study protocol), with ZioXT ECG patch monitor as the gold standard
Other arrhythmias | 1 year
  Incidence of Detection of other potentially clinically important non-AF arrhythmias: atrial tachycardia, pause >3 seconds, high-grade atrioventricular block (Mobitz type II or third-degree AV block), ventricular tachycardia, polymorphic ventricular tachycardia/ventricular fibrillation. ( within 12 months post-enrolment)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Healey, Principal Investigator — Population Health Research Institute
Locations (3):
- Canada (3):
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Health Centre, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] McIntyre WF, Vadakken ME, Connolly SJ, Mendoza PA, Lengyel AP, Rai AS, Latendresse NR, Grinvalds AJ, Ramasundarahettige C, Acosta JG, Um KJ, Roberts JD, Conen D, Wong JA, Devereaux PJ, Belley-Cote EP, Whitlock RP, Healey JS. Atrial Fibrillation Recurrence in Patients With Transient New-Onset Atrial Fibrillation Detected During Hospitalization for Noncardiac Surgery or Medical Illness : A Matched Cohort Study. Ann Intern Med. 2023 Oct;176(10):1299-1307. doi: 10.7326/M23-1411. Epub 2023 Oct 3. PMID 37782930